CLINICAL TRIAL: NCT01848548
Title: Superior Laryngeal Nerve Block For Airway Anesthesia Efficacy Study
Brief Title: Superior Laryngeal Nerve Block For Awake Endotracheal Intubation Study
Status: Terminated | Type: Observational
Why Stopped: Unable to continue recruit subjects
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: SLN Airway Trial
Record Dates: First submitted 2013-02-19; First posted 2013-05-07 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Awake Endotracheal Intubation; Difficult Intubation; Airway Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Assessment of Superior Laryngeal Nerve Block Technique
  Interventions: Procedure: Superior Laryngeal Nerve Block using the Thyrohyoid Membrane as an Anatomic Landmark

INTERVENTIONS:
Procedure: Superior Laryngeal Nerve Block using the Thyrohyoid Membrane as an Anatomic Landmark — The needle is introduced just lateral to midline above the thyroid notch in a slightly medial direction so as to enter the thyrohyoid membrane, and inserted about 1-1.5 cm. Three milliliters of 2% lidocaine is injected.

SUMMARY:
Awake tracheal intubation is the standard management for patients as risk for airway compromise. It is also commonly done in cases where there is significant cervical spine pathology i.e. cervical myelopathy or instability. The anesthetic technique used for the awake intubation is crucial to the patient's safety. One of the most important aspects of the anesthetic technique is airway anesthesia prior to placement of an endotracheal tube. The superior laryngeal nerve is responsible for mediating the cough reflex around the vocal cords. The investigators have developed an approach to reliably block the superior laryngeal nerve by injecting local anesthetic near the nerve in a unique approach. Injecting local anesthetic into or through the thyrohyoid membrane will effectively block the superior laryngeal nerve

ELIGIBILITY:
Inclusion Criteria

1. Patients between the ages of 18-80 requiring an awake intubation for endotracheal intubation.
2. Ability to speak and understand English

Exclusion Criteria

1. Allergy to lidocaine
2. Emergent operative case
3. Therapeutic anticoagulation
4. Mouth opening less than 2 cm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Scheduled Surgery Patients who require an awake intubation
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-04; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is to assess the efficacy of blocking the superior laryngeal nerve by using cough at the vocal cords on a 4 point scale | Immediate Perioperative period

SECONDARY OUTCOMES:
Time to placement of block | Immediate Perioperative Period

OTHER OUTCOMES:
During the intubation the lowest mean arterial blood pressure (MAP) | Immediate Perioperative Period
The lowest heart rate(HR) during intubation | Immediate Perioperative Period
The lowest respiratory rate during the intubation | Immediate Perioperative Period

CONTACTS AND LOCATIONS:
Overall Officials: Scott Miller, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States